CLINICAL TRIAL: NCT01958801
Title: Comparison Between Ultrasound-guided Supraclavicular and Interscalene Brachial Plexus Blocks in the Patients Undergoing Arthroscopic Shoulder Surgery
Brief Title: Clinical Efficacy of Supraclavicular Block for Arthroscopic Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, JongHae Kim, Assistant Professor, Daegu Catholic University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CR-13-033
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Horner's Syndrome
Keywords: Supraclavicular brachial plexus block; Interscalene brachial plexus block; Arthroscopic shoulder surgery
MeSH Terms: conditions — Horner Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interscalene block (Active Comparator): Interscalene block is performed under ultrasound guidance. Linear probe is placed on the ipsilateral interscalene groove visualizing the brachial plexus located between anterior and middle scalene muscles. Using in-plane technique, nerve stimulation needle is advanced into the brachial plexus sheath, into which 25 ml of 1.5% mepivacaine is injected.
  Interventions: Other: Interscalene block
- Supraclavicular block (Experimental): Supraclavicular block is performed under ultrasound guidance. Linear probe is placed on the ipsilateral supraclavicular fossa visualizing the brachial plexus located lateral to the subclavian artery. Using in-plane technique, nerve stimulation needle is advanced into the brachial plexus sheath, into which 25 ml of 1.5% mepivacaine is injected.
  Interventions: Other: Supraclavicular block

INTERVENTIONS:
Other: Supraclavicular block — Redirection of the needle is allowed when spread of local anesthetics does not surround the brachial plexus appropriately and involuntary movement of the forearm or hand is not necessary to confirm the correct placement of the needle.
  Arms: Supraclavicular block
Other: Interscalene block — Redirection of the needle is allowed when spread of local anesthetics does not surround the brachial plexus appropriately and involuntary movement of the forearm or hand is not necessary to confirm the correct placement of the needle.
  Arms: Interscalene block

SUMMARY:
The aim of this study is to compare the efficacy of supraclavicular and interscalene brachial plexus blocks in the patients undergoing arthroscopic shoulder surgery.

DETAILED DESCRIPTION:
This study aims to compare supraclavicular brachial plexus block to interscalene brachial plexus block with regard to degree of sensory and motor blockades, side effects and complications of the blocks, and frequency of intraoperative analgesics or antihypertensives use.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I-II
* Body mass index < 35 kg/m2

Exclusion Criteria:

* Neurologic deficits on the side to be blocked
* Infection or inflammation at the puncture site for brachial plexus block
* Psychiatric disorders
* Patient refusal
* Difficulty to communicate
* Coagulation deficiencies

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Degree of sensory blockade | 20 minutes after the end of local anesthetics injection
  Sensory blockade of the C5 to T1 dermatomes was assessed by rating the absence of cold sensation between 100 (intact sensation) and 0 (no sensation) with an alcohol swab.

SECONDARY OUTCOMES:
Degree of motor blockade | 20 minutes after the end of local anethetics injection
  Motor blockade was evaluated by elbow and wrist extension (radial nerve), finger abduction (ulnar nerve), wrist flexion (median nerve), and elbow flexion (musculocutaneous nerve). The muscle force was rated on a scale of 0 to 6 as follows (6: normal muscle force; 5: slightly reduced muscle force; 4: greatly reduced muscle force; 3: slightly impaired mobility; 2: greatly impaired mobility; 1: near complete paralysis; 0: complete paralysis).
Side effects | 20 minutes after the end of local anethetics injection
  Horner's syndrome (ptosis, miosis, anhidrosis) Subjective dyspnea Hoarseness
Frequency of intraoperative analgesics or antihypertensives use | At the end of the surgery
  Frequency of intraoperative use of opioids (fentanyl) or antihypertensives (hydralazine)

CONTACTS AND LOCATIONS:
Overall Officials: JongHae Kim, Master, Principal Investigator — Daegu Catholic University Medical Center
Locations (1):
- Daegu Catholic University Medical Center, Daegu, South Korea

REFERENCES:
- [Background] Liu SS, Gordon MA, Shaw PM, Wilfred S, Shetty T, Yadeau JT. A prospective clinical registry of ultrasound-guided regional anesthesia for ambulatory shoulder surgery. Anesth Analg. 2010 Sep;111(3):617-23. doi: 10.1213/ANE.0b013e3181ea5f5d. Epub 2010 Aug 4. PMID 20686013
- [Background] Conroy PH, Awad IT. Ultrasound-guided blocks for shoulder surgery. Curr Opin Anaesthesiol. 2011 Dec;24(6):638-43. doi: 10.1097/ACO.0b013e32834c155f. PMID 21934495